CLINICAL TRIAL: NCT01719406
Title: Randomized Control Pilot of a Behavior-based Exercise and Diet Intervention to Reduce Risk Factors for Gestational Diabetes Among Otherwise Healthy Pregnant Women.
Brief Title: The OHSU Pregnancy Exercise & Nutrition (PEN) Program
Acronym: PEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Linn Goldberg, Professor of Medicine, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: eIRB # 8895
Record Dates: First submitted 2012-10-29; First posted 2012-11-01 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2013-01

CONDITIONS: Gestational Diabetes
Keywords: Gestational diabetes; Exercise; Diet; Fruits; Vegetables; Whole grains; pregnancy weight
MeSH Terms: conditions — Diabetes, Gestational; Motor Activity | interventions — Methods; Nutritional Status; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention, behavioral lifestyle education (Experimental): Pregnant women will participate in 20 educational sessions designed to promote daily exercise, vegetable and fruit intake, maintain a diet that is relatively lower in fat and rich in whole grains.
  Interventions: Behavioral: Intervention, behavioral lifestyle education
- Control (No Intervention): Standard medical care

INTERVENTIONS:
Behavioral: Intervention, behavioral lifestyle education — Twenty interactive weekly sessions that are scripted curriculum and peer led.
  Other Names: Lifestyle; Nutrition; Exercise; Stress management
  Arms: Intervention, behavioral lifestyle education

SUMMARY:
Personal behaviors can influence development of Gestational Diabetes Mellitus (GDM), a condition that can adversely affect the pregnant woman, her developing fetus and future events for both. To reduce GDM risk, we will develop and implement an in-person team and web-based nutrition and exercise program for women, beginning in their first trimester. A scripted, peer-led, 20-week educational program, tailored for pregnant women working in teams (5 women/team), will be developed and implemented among pregnant employees and/or their spouses. Each weekly thirty minute session will focus on achieving 30-minutes of moderate daily physical activity with nutrition targets of five servings of fruits and vegetables, 3 servings of whole grains and lower fat food choices. Diet, exercise and lab assessments will occur before enrollment during the first trimester, each subsequent trimester and 12 weeks after delivery. In addition to exercise and diet survey results, we will assess fasting glucose, insulin, hemoglobin A1C levels, pregnancy weight gain, blood pressure, lipid and lipoprotein levels, pedometer records, weekly accelerometer data, each trimester and at 12 weeks post delivery, as well as gestational birth age, Apgar score, delivery mode and infant birth weight, and weekly health thermometer self-ratings during the assessment period.

ELIGIBILITY:
Inclusion Criteria: Healthy first trimester pregnant women -

Exclusion Criteria: hypertension, diabetes, known cardiopulmonary disease; orthopedic problems or other conditions that would prevent regular physical activity.

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Achieving 30 minutes of daily exercise, four or more times each week | 32 weeks
  Assessment of daily exercise (in minutes) during pregnancy and 12 weeks post pregnancy for the duration of the study.

SECONDARY OUTCOMES:
Eating 5 or more servings of vegetables and/or fruits each day | 32 weeks of the study
  Women will self-assess the number of servings of vegetables and fruits each day throughout the study.

OTHER OUTCOMES:
Pregnancy weight gain | 20 weeks
  Assess pregnancy weight gain, in which excessive weight gain is a risk factor for gestational diabetes.
HemoglobinA1C | Each trimester and 12-weeks post delivery
  Assessing the average plasma glucose concentration over longer time periods.

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States